CLINICAL TRIAL: NCT03952429
Title: SPIRA: Development of a Smartphone Based Intervention for the Prevention of Relapse in Alcohol Dependence
Brief Title: A Smartphone Based Intervention for the Prevention of Relapse in Alcohol Dependence
Acronym: SPIRA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Salus Klinik Lindow (Network)
Collaborators: University of Cambridge (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: SPIRA
Record Dates: First submitted 2019-05-10; First posted 2019-05-16 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Alcohol Dependence; Alcohol Abuse; Alcohol Use Disorder
Keywords: alcohol dependence; alcohol abuse; withdrawal
MeSH Terms: conditions — Alcoholism | interventions — Ethanol; Amyloid

STUDY DESIGN:
Intervention Model Description: This is a parallel study, participants will be randomised into 2 groups: one will be given the App with cognitive bias modification, whilst the other one will receive the app without the modification
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be notified there are 2 versions of the app and they will randomly be assigned to one of the 2 conditions, but will not know which one. Therapists giving the users input on how to use the app do not know in which condition the patient is either. Outcome (relapse rates) are assessed by interns and admin staff of the clinic who are independent from the study. The study investigators do not know the patients and only receive anonymized data on group and outcome variables.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Cognitive Bias App (Active Comparator): Participants will receive the Anti-Alcohol App with the Active Cognitive Bias modification, as well as participant diaries assessing alcohol consumption and several questionnaires.
  Interventions: Behavioral: Anti Alcohol App with Active Cognitive Bias
- Inactive Cognitive Bias Modification (Placebo Comparator): Participants will receive the Anti-Alcohol App with the Inactive Cognitive Bias Modification, as well as participant diaries assessing alcohol consumption and several questionnaires.
  Interventions: Behavioral: Inactive Cognitive Bias Modification

INTERVENTIONS:
Behavioral: Anti Alcohol App with Active Cognitive Bias — The active version includes an active form of cognitive bias modification, i.e. the user has to avoid alcohol stimuli 90% of the time, while they approach soft drinks 90% of the time.
  Arms: Active Cognitive Bias App
Behavioral: Inactive Cognitive Bias Modification — The control version includes an placebo form of cognitive bias modification, i.e. the users avoid and approach alcohol and softdrink stimuli for an equal number of trials.
  Arms: Inactive Cognitive Bias Modification

SUMMARY:
The rate of relapse following an inpatient alcohol rehabilitation program has been around 50% for a number of years. Offered treatments mainly focus on conscious and controllable aspects of behaviour, but research has found that much of the craving in addiction is guided by automatic processes, which are for a large part unconscious and poorly controlled by the individual. One way to influence these automatic processes is by applying cognitive bias modification, a cognitive-behavioural intervention that can be applied by a computer application. In alcohol addition, a common cognitive bias is the Alcohol-Approach bias. The Anti-Alcohol Training is a form of cognitive bias modification that was developed to reduce this approach bias and it has been shown to reduce the rates of relapse by 4-8%. A drawback of the training is that patients do not continue this at home after discharge. One way to increase accessibility is to offer the training in an app-game form.

In this study the investigators have developed a smartphone based training app that allows patients to more easily use the Anti-Alcohol training at home after discharge. The study aims to assess whether use of the app further reduces the alcohol bias and whether it can reduce yearly relapse rates.

DETAILED DESCRIPTION:
The rate of relapse following an inpatient alcohol rehabilitation program has been around 50% for a number of years, in spite of many initiatives to try and reduce relapse. One of the reasons could be that the offered treatments mainly focus on conscious and controllable aspects of behaviour. Recent research has however found that much of the craving in addiction is guided by automatic processes, which are for a large part unconscious and poorly controlled by the individual. Unsurprisingly, many attempts have therefore been made in addition research to reduce these automatic impulsive behaviour and improve the control processes.

One way to influence these automatic processes is by applying cognitive bias modification, a cognitive-behavioural intervention that can be applied by a computer application. In alcohol addition, a common cognitive bias is the Alcohol-Approach bias, the tendency to automatically approach alcohol. The Anti-Alcohol Training is a form of cognitive bias modification that was developed to reduce this approach bias. Studies have shows that this training can reduce the rates of relapse by 4-8%.

A drawback of the training is that patients often do not continue this at home after discharge, probably due to low motivation. One way to resolve this issue could be to offer the training in an App-game form, which would make it more accessible and inviting to continue using it after return home.

In this study the investigators have developed a smartphone based training app that allows patients to more easily use the Anti-Alcohol training at home after discharge. The study aims to assess whether alcohol dependent patients continue to use this app at home, whether the use of the app further reduces the alcohol bias, and finally whether it can reduce yearly relapse rates.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of Alcohol dependence / Alcohol Use disorder
* Taking part in alcohol rehabilitation program in Salus Clinic Lindow or being part of a self-help group

Exclusion Criteria:

* Visual or motor impairments that would affect the use of smartphones

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2019-05-23 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Relapse Rates | 3 months after care
  Relapse rates after leaving inpatient care, assessed through standard clinic follow-ups
App Usage | within 3 months after leaving care
  Number of times App training has been completed
Craving | after 5 training sessions of the app
  Craving for alcohol assessed in app, 5 point likert scale with alcohol images, OCDS

CONTACTS AND LOCATIONS:
Overall Officials: Prof Johannes Lindemeyer, Principal Investigator — Medizinische Hochschule Brandenburg Theodor Fontane
Locations (1):
- Salus Klinik Lindow, Lindow, Brandenburg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Anonymised participant data will be shared with the collaborators at Cambridge University
Supporting Information: Study Protocol, SAP, ICF, Analytic Code